CLINICAL TRIAL: NCT01755429
Title: A Research Study to Describe the Safety and Efficacy of Eculizumab in Japanese Patients With Atypical Hemolytic Uremic Syndrome (aHUS). An Assessment of Two Case Studies
Brief Title: To Characterize the Safety and Tolerability of Eculizumab in Two Japanese aHUS Patients
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C11-004J
Record Dates: First submitted 2012-12-04; First posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-02

CONDITIONS: ATYPICAL HEMOLYTIC UREMIC SYNDROME (AHUS)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol is intended to formally collect data on the treatment of aHUS with eculizumab in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and/or legal guardian must be willing and able to give written informed consent and id the patient is not an adult and able to read and write, the patient is willing to give written informed assent
2. Eculizumab treatment initiated as personal importation for aHUS in 201

Exclusion Criteria:

Not Applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The two identified Japanese patients with aHUS for which eculizumab treatment was initiated in 2011
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in platelet count from baseline | 26 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Shinshu University School of Medicine, Matsumoto
  - Tokyo Medical and Dental University, Tokyo